CLINICAL TRIAL: NCT02100176
Title: Multidisciplinary Intensive Rehabilitation Treatment and Rotigotine in the Early Stages of Parkinson's Disease: a Randomized Controlled Study.
Brief Title: MIRT and Rotigotine in the Early Stage of PD
Acronym: MIRT-RT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Other Study IDs: MIRT-RT; MIRT-RT (Other: Ospedale Generale di Zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson's Disease
Keywords: Rehabilitation treatment
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Rotigotine and MIRT: Group 1 - 20 Patients with PD (H&Y stages 1,5-2) in therapy only with Rotigotine will undergo a Multidisciplinary intensive rehabilitation treatment (MIRT).
  Interventions: Other: Multidisciplinary intensive rehabilitation treatment; Drug: Rotigotine
- Control group, only Rotigotine: Group 2 - 20 Patients with PD (H&Y stages 1,5-2)
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Other: Multidisciplinary intensive rehabilitation treatment — The first session comprises cardiovascular warm-up activities, relaxation exercises, muscle-stretching exercises, exercises to improve the range of motion of spinal, pelvic and scapular joints, exercises to improve the functionality of the abdominal muscles, and postural changes in supine position. The second session comprises exercises to improve balance and gait using a stabilometric platform with a visual cue and treadmill plus. The last session is a session of occupational therapy aimed to improve autonomy in daily living activities.
  Groups: Rotigotine and MIRT
Drug: Rotigotine — Rotigotine 2-8 mg/24 h
  Other Names: Dopamine agonist drug

SUMMARY:
To test whether a multidisciplinary intensive rehabilitation treatment (MIRT) slowed down the progression of the disease in Parkinson's disease (PD) "de novo" patients, all treated with Rotigotine, in a randomized controlled study with a 18 months follow-up.

DETAILED DESCRIPTION:
In the last years different rehabilitation treatments have been proposed to address specific motor deficits in Parkinson's disease. Nevertheless, the evidence of a possible neuroprotective action of exercise in PD has been obscured by the facts that all studies were performed in patients in different disease stages and under a variety of pharmacological treatments. Our objective is to test whether a multidisciplinary intensive rehabilitation treatment (MIRT) slowed down the progression of the disease in PD "de novo" patients, all treated with Rotigotine, in a randomized controlled study with a 18 months follow-up.

40 Patients at the initial stages of PD (H&Y stages 1,5-2) treated only with Rotigotine will be enrolled and randomly assigne into two groups. Patients in group 1 (20 subjects) will be undergone 2 MIRT cycle (at T0 and T3). MIRT consist of a 4-week cycle of physiotherapy that entailed three daily sessions 5 days a week (Frazzitta G. et al., Neurorehabilitation [30] 2012, 295-301). Patients in Group 2 (20 subjects) will continue with drug therapy alone.

For the group 1, Unified Parkinson's disease rating scale (UPDRS) II, UPDRS III, six-minute walking test (6MWT), Berg Balance Scale (BBS), Timed-up-and-go test (TUG), comfortable and fast gait speed, Self-assessment Parkinson's disease disability scale and L-dopa equivalents will be assessed at Baseline T0, T1 (discharge after the first MIRT cycle), T2 (control at 6 months after discharge), T3 (hospitalization for second MIRT cycle), T4 (discharge after the second MIRT cycle) and T5 (end of the protocol, 18 months); For the group 2, UPDRS II, UPDRS III, six-minute walking test (6MWT), Berg Balance Scale (BBS), Timed-up-and-go test (TUG), confortable and fast gait speed, Self-assessment Parkinson's disease disability scale and L-dopa equivalents will be assessed at Baseline T0, T1 (check-up at 6 months), T2 (check-up at 12 months), T3 (check-up at 18 months).

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease according to Gelb et al., ability to walk without any physical assistance, no cognitive impairment (MMSE score > 26), no comorbidity unrelated to Parkinson's disease, no vestibular/visual dysfunction limiting locomotor or balance.

Exclusion Criteria:

* Atypical Parkinsonisms, cognitive impairment (MMSE < 26), other comorbidities not related to PD, vestibular/visual dysfunction limiting locomotor or balance.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease "de novo" Patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
UPDRS total score | 18 Months
  Unified Parkinson's Disease Rating Scale total score

SECONDARY OUTCOMES:
UPDRS II | 18 Months
  Unified Parkinson's disease Rating Scale II
UPDRS III | 18 Months
  Unified Parkinson's disease Rating Scale
6MWT | 18 Months
  Six Minutes Walking Test
BBS | 18 Months
  Berg Balance Scale
TUG | 18 Months
  Time up and go test
CGS and FGS | 18 Months
  Comfortable and fast gait speed
SPDDS | 18 Months
  Self-Assessment Parkinson's Disease Disability Scale

OTHER OUTCOMES:
L Dopa | 18 Months
  levo-dopa equivalent dosage

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti 22015 - CO, Italy
Locations (2):
- Italy (2):
  - Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona, Como
  - Riabilitazione Neuromotoria, Istituto Scientifico di Montescano, Montescano, Pavia